CLINICAL TRIAL: NCT03544632
Title: A Phase II, Dose-escalation, Open-label Study Evaluating the Safety and Efficacy of Permanently-placed Acellular Adipose Tissue (AAT) in Human Subjects With Modest Soft Tissue Defects of the Trunk
Brief Title: Acellular Adipose Tissue (AAT) for Soft Tissue Reconstruction
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency); Armed Forces Institute of Regenerative Medicine (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00155003
Record Dates: First submitted 2018-04-25; First posted 2018-06-04 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Soft Tissue Injuries; Trauma
Keywords: adipose-derived extracellular matrix (ECM); acellular adipose tissue (AAT)
MeSH Terms: conditions — Soft Tissue Injuries; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Acellular Adipose Tissue (AAT) (Experimental): This open-label, phase II, dose-escalation study will be conducted in human subjects seeking repair of modest (approx. 5-30cc) soft tissue defects of the trunk (n=15). All participants will be treated via permanent injection of the study intervention (AAT injection) to restore the defect's contour. All study data will be collected in Case Report Forms (CRFs) and entered into a customized study database, created and maintained in HIPAA-compliant Research Electronic Data Capture (REDCap) software (14).
  Interventions: Drug: Acellular Adipose Tissue (AAT)

INTERVENTIONS:
Drug: Acellular Adipose Tissue (AAT) — Participants (n=15) will be administered between 5cc and 20cc of AAT, depending on their assigned treatment group, via sterile subcutaneous injection into the target defect. The injection is intended to be permanent. After the 3-month study follow-up visit, participants will have the option to undergo additional AAT injection (up to 20cc per treatment) in order to fully correct the defect. Total injected AAT volume per patient will not exceed 40cc. Additional injection is dependent upon study- and patient-specific adverse / unanticipated events to date.
  Each vial contains a 2 milliliter (mL) dose of the injectable AAT. This volume is similar to other commonly used injectable filler materials intended for soft tissue correction.

SUMMARY:
Although other methods (e.g., autologous fat transfer, dermal-/collagen-based fillers) for soft tissue reconstruction exist, each has distinct disadvantages leaving room for improvement in this treatment area. Investigators in the Elisseeff Laboratory (Johns Hopkins University Department of Biomedical Engineering) have recently generated a novel tissue-derived material to create instructive matrices for soft tissue reconstruction called Acellular Adipose Tissue (AAT). This material takes advantage of the inherent bioactivity and unique mechanical properties of subcutaneous adipose tissue. Investigators' preclinical data suggest that AAT is safe for use in small and large animals; investigators' clinical (Phase I) data suggest that AAT is safe for use in humans. These data indicate that a Phase II, dose-escalation study of AAT's safety and efficacy in human subjects is warranted.

DETAILED DESCRIPTION:
Soft tissue volume loss acquired through trauma, congenital malformation or comorbid conditions (i.e., HIV/AIDS) is a common and sometimes devastating problem. Traditional therapies include local tissue transfer, allograft placement, and complex scar revision techniques. Recently, autologous fat transfer has become one of the most commonly employed techniques for improving soft tissue contour deformity particularly for the correction of breast and body defects. While the results from this procedure continue to improve, it requires an additional procedure to harvest fat tissue from the abdomen, thigh or flank leading to donor site morbidity. Clinically, volume loss following autologous fat transfer has been reported to be between 40-60% and usually occurs within the first 4-6 months. Regrafting is often needed and implanted adipose tissue frequently leads to post-operative calcifications. For these reasons, a predictable, "off-the-shelf" material that retains the mechanical and biological properties of adipose tissue would be ideal for the reconstruction of smaller soft tissue defects and soft tissue augmentation.

Investigators in the Elisseeff Laboratory (Johns Hopkins University Department of Biomedical Engineering) generated a novel tissue-derived material to create instructive matrices for soft tissue reconstruction [Acellular Adipose Tissue (AAT)]. In 2016, investigators conducted a Phase 1, open-label, clinical trial of AAT in healthy volunteers who planned to have elective surgery for the removal of redundant tissue (n=8). Overall, AAT demonstrated satisfactory safety results. No participants experienced serious adverse events (SAEs) or unanticipated adverse events (AEs) related to the study, or exited the study due to AEs. All AEs noted were expected and mild, including redness, bruising, textural changes, hyperpigmentation and tenderness at the injection site. Many other adverse events commonly associated with injections were not observed in any participant throughout the study (i.e., scarring, ulceration, scabbing, purpura, oozing, crusting, blanching, blistering, edema or abrasions). These data indicate that conducting a phase II, dose-escalation, safety and efficacy study in humans is warranted. Based on investigators' experience, investigators hypothesize that AAT will be safe and maintain its volume up to 6 months when injected subcutaneously to restore 5-20cc defects in human soft tissue.

ELIGIBILITY:
Inclusion Criteria:

Men and women aged 18-65 years with at least one modest (5-30cc) soft tissue defect on the trunk and

* Willingness to wait up to 6 months to participate in the study (depending on defect size and enrollment-to-date).
* Consent to photography for research purposes.
* Willingness to follow study requirements.
* Ability to give informed consent.
* Willingness to perform follow up visits for 12 months (+/- 30 days).
* Willingness to undergo complete blood count (CBC) with Differential and Serum Chemistry.

For Men and Women of reproductive potential: Willingness to use approved methods of birth control or abstain from sexual intercourse from screening until 6 months post-AAT injection.

* Definition of non-childbearing potential for Women: amenorrhea (previous 12 months) or surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy).
* Definition of non-reproductive potential for Men: confirmed surgically sterile (vasectomy >3 months prior to screening).

Exclusion Criteria:

Use of AAT in patients exhibiting autoimmune connective tissue disease is not recommended. When applied properly, AAT has been shown to support the migration of host cells from the surrounding tissue. Therefore, this study will exclude patients with conditions that could inhibit migration of host cells including, but not limited to, the following:

* Fever (oral temperature >99º F at time of screening)
* Insulin dependent diabetes
* Low vascularity of the tissue intended for elective excision
* Local or Systemic Infection
* Mechanical Trauma
* Poor nutrition or general medical condition
* Dehiscence and/or necrosis due to poor revascularization
* Specific or nonspecific immune response to some component of the AAT material
* Infected or nonvascular surgical sites
* Known cancer or receiving treatment for cancer

Also:

* Pregnant or Lactating females
* Inability to cooperate with and/or comprehend post-operative instructions
* Inability to speak or read English
* Known allergy or sensitivity to Streptomycin or Amphotericin B
* Any other reason the study physicians judge would be a contraindication for receiving AAT injections

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2018-06-21 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
AAT efficacy for soft-tissue reconstruction - Volume Retention | 6 months post-final injection
  Volume retention documented by pre-to-post injection volumetric changes as detected by 3-dimensional photography
AAT efficacy for soft-tissue reconstruction - blinded assessors | 6 months post-final injection
  Assessments to determine aesthetic appearance of defects documented by blinded assessors rating defect sites using the Global Aesthetic Improvement Scale (GAIS). 5 point scale ranging from 1 to 5 with 5 = The appearance has worsened compared with the original condition and 1 = Excellent corrective results
AAT efficacy for soft-tissue reconstruction - patient-reported | 6 months post-final injection
  Post-injection assessment to determine aesthetic outcome documented by patient-reported satisfaction with the repair

SECONDARY OUTCOMES:
Histopathological analysis of explanted implants | up to 12 months post-injection
  Histopathology will be performed on core needle biopsy samples collected at 3, 6, 9, and 12 months post-injection and will be done using the following: H&E staining to assess (1) native cellular infiltration of the implant, (2) location of implant relative to dermis/subdermis, (3) inflammatory response to implant, and (4) presence of fibrosis
Physician Ease of Use Assessments | up to 12 months post-injection
  Physician ease of use will be measured through the completion of self-administered surveys by the study surgeon.
Participant Comfort Surveys | up to 12 months post-injection
  Participant comfort will be measured through the completion of self-administered surveys by the participant.

CONTACTS AND LOCATIONS:
Overall Officials: Damon Cooney, MD, PhD, Principal Investigator — The Department of Plastic and Reconstructive Surgery, Johns Hopkins University School of Medicine
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bucky LP, Percec I. The science of autologous fat grafting: views on current and future approaches to neoadipogenesis. Aesthet Surg J. 2008 May-Jun;28(3):313-21; quiz 322-4. doi: 10.1016/j.asj.2008.02.004. PMID 19083543
- [Background] Wan DC, Lim AT, Longaker MT. Craniofacial autologous fat transfer. J Craniofac Surg. 2009 Mar;20(2):273-4. doi: 10.1097/SCS.0b013e31819921d3. No abstract available. PMID 19305242
- [Background] Cordeiro PG. Breast reconstruction after surgery for breast cancer. N Engl J Med. 2008 Oct 9;359(15):1590-601. doi: 10.1056/NEJMct0802899. No abstract available. PMID 18843123
- [Background] Rosson GD, Magarakis M, Shridharani SM, Stapleton SM, Jacobs LK, Manahan MA, Flores JI. A review of the surgical management of breast cancer: plastic reconstructive techniques and timing implications. Ann Surg Oncol. 2010 Jul;17(7):1890-900. doi: 10.1245/s10434-010-0913-7. Epub 2010 Mar 9. PMID 20217253
- [Background] Pulagam SR, Poulton T, Mamounas EP. Long-term clinical and radiologic results with autologous fat transplantation for breast augmentation: case reports and review of the literature. Breast J. 2006 Jan-Feb;12(1):63-5. doi: 10.1111/j.1075-122X.2006.00188.x. PMID 16409589
- [Background] Cheng MH, Uriel S, Moya ML, Francis-Sedlak M, Wang R, Huang JJ, Chang SY, Brey EM. Dermis-derived hydrogels support adipogenesis in vivo. J Biomed Mater Res A. 2010 Mar 1;92(3):852-8. doi: 10.1002/jbm.a.32410. PMID 19280638
- [Background] Uriel S, Huang JJ, Moya ML, Francis ME, Wang R, Chang SY, Cheng MH, Brey EM. The role of adipose protein derived hydrogels in adipogenesis. Biomaterials. 2008 Sep;29(27):3712-3719. doi: 10.1016/j.biomaterials.2008.05.028. Epub 2008 Jun 24. PMID 18571717
- [Background] Wu I, Nahas Z, Kimmerling KA, Rosson GD, Elisseeff JH. An injectable adipose matrix for soft-tissue reconstruction. Plast Reconstr Surg. 2012 Jun;129(6):1247-1257. doi: 10.1097/PRS.0b013e31824ec3dc. PMID 22327888
- See also: Safety Study of Acellular Adipose Tissue for Soft Tissue Reconstruction — https://clinicaltrials.gov/ct2/show/NCT02817984